CLINICAL TRIAL: NCT01673919
Title: Long-term, Interventional, Open Label Extension Study Evaluating the Safety of Tocilizumab Treatment in Patients With Polyarticular-course Juvenile Idiopathic Arthritis From France Who Completed the Global, Multinational Trial (WA19977)
Brief Title: A Long-Term Extension Study of RoActemra/Actemra (Tocilizumab) in Patients With Juvenile Idiopathic Arthritis From France Who Completed WA19977 Core Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28166; 2011-005515-90 (EudraCT Number)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- RoActemra/Actemra (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, 104 weeks

SUMMARY:
This long-term, open-label extension study will evaluate the safety of RoActemra/Actemra (tocilizumab) in patients with polyarticular-course juvenile idiopathic arthritis who completed the WA19977 core study. Patients will continue to receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks. Anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed visit 33 (week 104) of WA19977 study and who may benefit from study drug treatment according to the investigator's assessment
* Patients have to receive the first RoActemra/Actemra infusion in this study at the Week 8 visit at the latest
* Females of child-bearing potential and males with female partners of child-bearing potential must agree to use effective contraception as defined by protocol

Exclusion Criteria:

* Patients with, according to investigator judgment, not satisfactory benefit from RoActemra/Actemra therapy within WA19977
* Treatment with any investigational agent since the last administration of study drug in the core study WA19977
* Patient developed any other autoimmune rheumatic disease or overlap syndrome other than the permitted polyarticular-course Juvenile Idiopathic Arthritis (JIA) subsets: rheumatoid factor positive or negative JIA or extended oligoarticular JIA
* Patient is pregnant , lactating, or intending to become pregnant during the study and up to 12 weeks after the last administration of study drug
* Any significant concomitant disease or medical or surgical condition
* History of significant allergic or infusion reactions to prior biologic therapy
* Currently active primary or secondary immunodeficiency
* Any infections with contraindications to RoActemra/Actemra therapy according to investigator judgment
* Inadequate hepatic, renal or bone marrow function

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- France (3):
  - Le Kremlin-Bicêtre
  - Montpellier
  - Paris

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of seven participants who completed the core study WA19977 were enrolled in this extension study conducted from 13 February 2012 to 15 January 2014 at four centers in France.
Groups:
- Tocilizumab (8 mg/kg): Eligible participants received tocilizumab (TCZ) 8 milligram/kilogram (mg/kg) intravenously every 4 weeks up to 104 weeks or until TCZ was commercially available for polyarticular-course Juvenile Idiopathic Arthritis (pcJIA) in France, whichever came first.
Period: Overall Study
Arm/Group | Tocilizumab (8 mg/kg)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all the participants who had at least one efficacy assessment.
Groups:
- Tocilizumab (8 mg/kg): Eligible participants received TCZ 8 mg/kg intravenously every 4 weeks up to 104 weeks or until TCZ was commercially available for pcJIA in France, whichever came first.
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
Age, Customized [Number; unit: participants]
  2 to 11 years | 3
  12 to 17 years | 2
  18 to 64 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Any AEs | 7
  Any SAEs | 0

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. The AEs of special interests included gingival bleeding, tooth abscess, acarodermatitis, ear infection, gastroenteritis, herpes zoster ophthalmic, lice infestation, nasopharyngitis, oral fungal infection, oral herpes, pharyngitis, rhinitis, sinusitis, tonsillitis, tracheitis, tracheobronchitis, urinary tract infection, menorrhagia, asthma, epistaxis, and hematoma.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Gingival bleeding | 2
  Tooth abscess | 2
  Acarodermatitis | 1
  Ear infection | 1
  Gastroenteritis | 1
  Herpes zoster ophthalmic | 1
  Lice infestation | 1
  Nasopharyngitis | 1
  Oral fungal infection | 1
  Oral herpes | 1
  Pharyngitis | 1
  Rhinitis | 1
  Sinusitis | 1
  Tonsillitis | 1
  Tracheitis | 1
  Tracheobronchitis | 1
  Urinary tract infection | 1
  Menorrhagia | 1
  Asthma | 1
  Epistaxis | 1
  Hematoma | 1

3. Primary Outcome: Number of Participants With Adverse Events Related to Tocilizumab
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. Relatedness of any AEs was reported as possibly related, probably related, or remotely related to TCZ.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  AEs possibly related to TCZ | 5
  AEs probably related to TCZ | 2
  AEs remotely related to TCZ | 1

4. Secondary Outcome: Mean Exposure to Study Treatment
Description: Participants received TCZ for Week 104 or when TCZ was commercially available for pcJIA participants, whichever comes first in France. The mean TCZ exposure (time from first to last administration) was reported.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
Months | 17.08 (1.55)

5. Secondary Outcome: Mean Duration of Study Follow-Up
Description: The participants were followed-up from Day 1 to last visit date (approximately 2 years). Mean time for which participants were followed up in the study was reported.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
Months | 21.08 (1.64)

6. Secondary Outcome: Number of Participants With AEs Leading to TCZ Modification, AEs Leading to Death, Anaphylaxis or Serious Hypersensitivity and Deaths
Description: Number of participants with AEs leading to TCZ modification, AEs leading to death, anaphylaxis or serious hypersensitivity, and deaths were reported.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  AEs leading to TCZ modification | 2
  AEs leading to death | 0
  Anaphylaxis or serious hypersensitivity | 0
  Death | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Clinically significant abnormal parameters included eosinophil count, alanine aminotransferase, total bilirubin, and protein and blood in urine. Number of participants with these abnormal lab parameters was reported.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Eosinophil count | 1
  Alanine aminotransferase | 1
  Total bilirubin | 1
  Protein and blood in urine | 2

8. Secondary Outcome: Number of Participants With Abnormality in Physical Examinations
Description: Participants with abnormal physical examinations of ear, nose and throat (asthma); extremities (synovitis, sequelae with flexion of the 5th right proximal interphalangeal joint, hallux valgus, deviations of metatarsophalangeal joints, and callus under metatarsal head); lung (mild bronchospasm); skin (vitiligo and hematoma, fatty subcutaneous infiltration on the neck, cutaneous eruption, and scalp pediculosis); and musculoskeletal system (discomfort in right hip) were reported.
Time Frame: Approximately 2 years
Population: Safety population included all participants who received at least a single dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Ear, nose and throat | 1
  Extremities | 1
  Lung | 1
  Musculoskeletal system | 1
  Skin | 3

9. Secondary Outcome: Number of Participants With Juvenile Idiopathic Arthritis American College of Rheumatology Response 50/70
Description: The Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) is comprised of six components: Maximum number of joints with active arthritis; Number of joints with limitation of movement; Erythrocyte Sedimentation Rate (ESR) and/or C-reactive Protein (CRP); Childhood Health Assessment Questionnaire-Disease Index (CHAQ-DI) graded on 4-point scales [0 = without any difficulty and 3 = unable to do] of 30 items grouped into 8 domains of physical function; Physician's global assessment of disease activity and Participant's global assessment of overall well-being (both assessed on a 0 to 100 mm Visual Analogue Scale [VAS], where score 0 = inactive arthritis and 100 = very active arthritis). A JIA ACR50/70 response is defined as improvement in at least three of the six core components by at least 50 percent (%), or 70%, respectively and no more than one of the remaining core components worsening by more than 30%.
Time Frame: Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: The ITT population included all participants who had at least one efficacy assessment. Number (n) = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 6
participants
  JIA ACR50, Week 12 (n = 5): number analyzed (Participants) | 5
  JIA ACR50, Week 12 (n = 5) | 1
  JIA ACR50, Week 24 (n = 5): number analyzed (Participants) | 5
  JIA ACR50, Week 24 (n = 5) | 2
  JIA ACR50, Week 36 (n = 6) | 1
  JIA ACR50, Week 48 (n = 5): number analyzed (Participants) | 5
  JIA ACR50, Week 48 (n = 5) | 1
  JIA ACR50, Week 60 (n = 5): number analyzed (Participants) | 5
  JIA ACR50, Week 60 (n = 5) | 0
  JIA ACR50, Week 72 (n = 2): number analyzed (Participants) | 2
  JIA ACR50, Week 72 (n = 2) | 0
  JIA ACR50, Week 84 (n = 1): number analyzed (Participants) | 1
  JIA ACR50, Week 84 (n = 1) | 1
  JIA ACR50, Week 108 (n = 6) | 2
  JIA ACR70, Week 12 (n = 5): number analyzed (Participants) | 5
  JIA ACR70, Week 12 (n = 5) | 4
  JIA ACR70, Week 24 (n = 5): number analyzed (Participants) | 5
  JIA ACR70, Week 24 (n = 5) | 3
  JIA ACR70, Week 36 (n = 6) | 5
  JIA ACR70, Week 48 (n = 5): number analyzed (Participants) | 5
  JIA ACR70, Week 48 (n = 5) | 4
  JIA ACR70, Week 60 (n = 5): number analyzed (Participants) | 5
  JIA ACR70, Week 60 (n = 5) | 5
  JIA ACR70, Week 72 (n = 2): number analyzed (Participants) | 2
  JIA ACR70, Week 72 (n = 2) | 2
  JIA ACR70, Week 84 (n = 1): number analyzed (Participants) | 1
  JIA ACR70, Week 84 (n = 1) | 0
  JIA ACR70, Week 108 (n = 6) | 4

10. Secondary Outcome: Number of Participants With Inactive Disease
Description: Inactive disease was defined as: 1) No joints with active arthritis (no swollen, painful and lack of motion joints), 2) No fever, rash, serositis, splenomegaly, or generalized lymphadenopathy attributable to JIA, 3) No active uveitis, 4) ESR and/or CRP within normal range, and 5) No disease activity according to Physician's global assessment of disease activity (<= 10 millimeters [mm] on a VAS). The participant's treating physician provided a rating of the participant's arthritis disease activity on a 0 to 100 mm horizontal scale where score 0 represented 'arthritis inactive' (i.e., symptom-free and no arthritis symptoms) and score 100 represented 'arthritis very active'.
Time Frame: Weeks 24, 36, 48, 72, and 108
Population: The ITT population included all participants who had at least one efficacy assessment. n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Week 24 (n = 6): number analyzed (Participants) | 6
  Week 24 (n = 6) | 1
  Week 36 (n = 7) | 1
  Week 48 (n = 6): number analyzed (Participants) | 6
  Week 48 (n = 6) | 1
  Week 72 (n = 4): number analyzed (Participants) | 4
  Week 72 (n = 4) | 1
  Week 108 (n = 7) | 1

11. Secondary Outcome: Number of Participants Achieving Clinical Remission
Description: Clinical remission was defined as inactive disease observed for at least 6 continuous months. Clinical remission was defined as per medication uptake as: Level 1 (clinical remission on medication), Level 2 (clinical remission off oral corticosteroid medication [still on TCZ]), Level 3 (clinical remission off both oral corticosteroid and methotrexate medication [still on TCZ]), and Level 4 (clinical remission off all anti-inflammatory medications [still on TCZ]). Number of participants at each clinical remission level was reported.
Time Frame: Weeks 24, 36, 48, 72, and 108
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Week 24, Remission level 1 (n = 7) | 1
  Week 36, Remission level 1 (n = 6): number analyzed (Participants) | 6
  Week 36, Remission level 1 (n = 6) | 5
  Week 48, Remission level 1 (n = 6): number analyzed (Participants) | 6
  Week 48, Remission level 1 (n = 6) | 1
  Week 72, Remission level 1 (n = 4): number analyzed (Participants) | 4
  Week 72, Remission level 1 (n = 4) | 1
  Week 108, Remission level 1 (n = 7) | 1

12. Secondary Outcome: Number of Participants With a Minimally Important Improvement in the Childhood Health Assessment Questionnaire-Disability Index
Description: The CHAQ-DI included questions on dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. The disability index (DI) of the original CHAQ was graded on 4-point categorical scales of 30 items grouped into 8 domains of physical function. The highest scoring item in each domain determined the score for that domain. The score for the disability index was the mean of domain scores ranging from 0 to 3 (0 = without any difficulty and 3 = unable to do) with higher scores meaning higher disability. Minimally important improvement in CHAQ-DI was defined as a change from baseline of WA19977 core study (Day 1/Visit 1) >=0.13 at each visit.
Time Frame: Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: The ITT population included all the participants who had at least one efficacy assessment. n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: participants
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
participants
  Week 12 (n=7) | 5
  Week 24 (n=7) | 5
  Week 36 (n=7) | 6
  Week 48 (n=7) | 5
  Week 60 (n=7) | 6
  Week 72 (n=3): number analyzed (Participants) | 3
  Week 72 (n=3) | 2
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 0
  Week 108 (n=7) | 6

13. Secondary Outcome: Number of Joints With Limitation of Motion
Description: The most frequent symptom reported by most participants was a limitation of motion (LOM) of joints and it was determined by physical examination. The mean joints with limitation of motion were reported.
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
joints
  Day 1 (n=7) | 11.4 (14.3)
  Week 12 (n=7) | 9.4 (11.9)
  Week 24 (n=6): number analyzed (Participants) | 6
  Week 24 (n=6) | 6.7 (8.4)
  Week 36 (n=7) | 8.1 (9.5)
  Week 48 (n=7) | 8.6 (10.5)
  Week 60 (n=7) | 10.3 (14.8)
  Week 72 (n=4): number analyzed (Participants) | 4
  Week 72 (n=4) | 8.5 (16.3)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 31.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 10.6 (13.4)

14. Secondary Outcome: Number of Joints With Active Range of Motion
Description: The active range of motion joints was counted by physical examination and mean joints was reported.
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
joints
  Day 1 (n=7) | 2.3 (2.5)
  Week 12 (n=7) | 1.4 (2.3)
  Week 24 (n=6): number analyzed (Participants) | 6
  Week 24 (n=6) | 2.2 (2.2)
  Week 36 (n=7) | 1.3 (1.8)
  Week 48 (n=7) | 2.0 (1.9)
  Week 60 (n=7) | 2.0 (2.2)
  Week 72 (n=4): number analyzed (Participants) | 4
  Week 72 (n=4) | 0.3 (0.5)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 0.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 1.1 (1.2)

15. Secondary Outcome: Number of Swollen Joints
Description: The swollen joints was counted by physical examination and mean swollen joints were reported.
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
joints
  Day 1 (n=7) | 1.6 (2.1)
  Week 12 (n=7) | 1.0 (2.2)
  Week 24 (n=6): number analyzed (Participants) | 6
  Week 24 (n=6) | 1.0 (1.7)
  Week 36 (n=7) | 0.9 (1.5)
  Week 48 (n=7) | 1.9 (1.8)
  Week 60 (n=7) | 1.7 (2.2)
  Week 72 (n=4): number analyzed (Participants) | 4
  Week 72 (n=4) | 0.3 (0.5)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 0.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 0.7 (1.3)

16. Secondary Outcome: Number of Painful Joints
Description: The painful joints were counted by physical examination and mean painful joints was reported.
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
joints
  Day 1 (n=7) | 1.9 (2.3)
  Week 12 (n=7) | 0.6 (0.8)
  Week 24 (n=6): number analyzed (Participants) | 6
  Week 24 (n=6) | 2.0 (2.8)
  Week 36 (n=7) | 0.7 (1.0)
  Week 48 (n=7) | 0.9 (1.1)
  Week 60 (n=7) | 0.7 (1.0)
  Week 72 (n=4): number analyzed (Participants) | 4
  Week 72 (n=4) | 0.5 (1.0)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 0.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 2.0 (4.0)

17. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: The Physician's global assessment of disease activity was recorded on a 0 to 100 mm horizontal VAS where score 0 represented 'arthritis inactive' (i.e., symptom-free and no arthritis symptoms) and score 100 represented 'arthritis very active' (higher score indicate worsening of disease).
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
millimeter (mm)
  Day 1 (n=7) | 8.6 (7.7)
  Week 12 (n=6): number analyzed (Participants) | 6
  Week 12 (n=6) | 4.2 (6.4)
  Week 24 (n=7) | 9.3 (12.2)
  Week 36 (n=7) | 6.7 (6.9)
  Week 48 (n=7) | 3.7 (3.6)
  Week 60 (n=7) | 4.0 (3.4)
  Week 72 (n=4): number analyzed (Participants) | 4
  Week 72 (n=4) | 2.8 (4.3)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 4.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 6.6 (7.1)

18. Secondary Outcome: Parent/Patient's Global Assessment of Disease Activity
Description: Parent/patient global assessment of disease activity was performed using 0 to 100 mm VAS, and higher the score of VAS, worse the disease status (0= absence of activity or sign or symptom; 100= maximal activity or signs or symptoms). No disease activity was defined as VAS <=10 mm.
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
mm
  Day 1 (n=7) | 14.9 (27.5)
  Week 12 (n=7) | 8.0 (12.2)
  Week 24 (n=7) | 12.7 (23.3)
  Week 36 (n=7) | 3.9 (6.8)
  Week 48 (n=7) | 10.1 (17.4)
  Week 60 (n=7) | 7.4 (8.3)
  Week 72 (n=3): number analyzed (Participants) | 3
  Week 72 (n=3) | 0.3 (0.6)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 73.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 12.1 (17.8)

19. Secondary Outcome: Parent/Patient's Discomfort Index (Pain)
Description: Participants or parents rated participant's pain by placing a horizontal line on a VAS of 0 (no pain) - 100 mm (unbearable pain). To describe the pain, a cut-off at 10 mm was used, and VAS <10 mm was defined as no pain.
Time Frame: Baseline (Day 1), Weeks 12, 24, 36, 48, 60, 72, 84, and 108
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab (8 mg/kg)
Number analyzed (Participants) | 7
mm
  Day 1 (n=7) | 15.0 (27.2)
  Week 12 (n=7) | 5.6 (7.7)
  Week 24 (n=7) | 7.7 (11.1)
  Week 36 (n=7) | 3.0 (3.1)
  Week 48 (n=7) | 12.9 (18.5)
  Week 60 (n=7) | 6.4 (7.3)
  Week 72 (n=3): number analyzed (Participants) | 3
  Week 72 (n=3) | 0.7 (0.6)
  Week 84 (n=1): number analyzed (Participants) | 1
  Week 84 (n=1) | 51.0 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  Week 108 (n=7) | 5.1 (9.0)

ADVERSE EVENTS:
Time Frame: Approximately 2 years
Description: Safety population included all participants who received at least a single dose of study drug.
Arm/Group | Tocilizumab (8 mg/kg)
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (8 mg/kg) (N=7)
Neutropenia (Blood and lymphatic system disorders) | 2
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Vaccination site pain (General disorders) | 1
Allergy to arthropod bite (Immune system disorders) | 1
Tooth abscess (Infections and infestations) | 2
Acarodermatitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Lice infestation (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Bite (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Curetting of chalazion (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.